CLINICAL TRIAL: NCT05843630
Title: Development and Validation of an Individualized Nomogram to Differentiate Uncomplicated From Complicated Acute Appendicitis in Adults: a Multicenter Study
Brief Title: Radiomic Modeling in Differentiating Uncomplicated From Complicated Acute Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kecheng Zhang (Other)
Responsible Party: Sponsor-Investigator, Kecheng Zhang, Department of General Surgery, Chinese PLA General Hospital First Medical Center, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: PLAGH202304
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Acute Appendicitis
Keywords: acute appendicitis; diagnosis; nomogram
MeSH Terms: conditions — Appendicitis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: Model construction based on training cohort
  Interventions: Diagnostic Test: without
- Validation cohort 1: Model validation in an independent validation cohort 1
  Interventions: Diagnostic Test: without
- Validation cohort 2: Model validation in an independent validation cohort 2
  Interventions: Diagnostic Test: without

INTERVENTIONS:
Diagnostic Test: without — without

SUMMARY:
Non-operative management (NOM) with antibiotics may be a safe alternative to surgery for uncomplicated appendicitis, but preoperative differentiation between uncomplicated and complicated appendicitis is challenging. The study aimed to develop a clinical-radiomics nomogram to distinguish uncomplicated from complicated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as acute appendicitis after appendectomy between January 2021 and December 2022.

Exclusion Criteria:

* age less than 18 years (no upper age limit);
* without CT examination within a week before surgery;
* difficult to outline the contours of the appendix due to inflammatory exudate;
* lack of clinical information.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults with pathologically diagnosed as acute appendicitis after appendectomy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-06-03 (Estimated); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of clinical-radiomic model for differentiating complicated from uncomplicated appendicitis | January 2021 to December 2022
  ROC curve will be plotted and the area under ROC curve will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Kecheng Zhang, Principal Investigator — Senior Department of General Surgery, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital First Medical Center, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided